CLINICAL TRIAL: NCT02589795
Title: A Phase I Clinical Trial to Assess the Safety and Immunogenicity of HIV DNA-C CN54ENV Immunisations Administered Via the IM and ID Methods With and Without Electroporation Followed by Boosting With Recombinant HIV CN54gp140 in Healthy Male and Female Volunteers
Brief Title: Safety and Immunogenicity of HIV DNA-C CN54ENV and Recombinant HIV CN54gp140 Vaccines in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CUTHIVAC002
Record Dates: First submitted 2015-10-21; First posted 2015-10-28 (Estimated); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: HIV
Keywords: safety; immunogenicity; HIV vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: ID/EP + IM (Experimental): 0.6 mg DNA-C CN54ENV, intradermally with electroporation, at Weeks 0, 4 and 8. 2 mg DNA-C CN54ENV, intramuscularly without electroporation, at Weeks 0, 4 and 8.
  50 µg CN54gp140, intradermally without electroporation, at Week 20.
  Interventions: Biological: DNA-C CN54ENV; Biological: CN54gp140; Device: Trigrid Delivery System - Intradermal
- Group 2: ID + IM/EP (Experimental): 0.6 mg DNA-C CN54ENV, intradermally without electroporation, at Weeks 0, 4 and 8.
  2 mg DNA-C CN54ENV, intramuscularly with electroporation, at Weeks 0, 4 and 8. 50 µg CN54gp140, intradermally without electroporation, at Week 20.
  Interventions: Biological: DNA-C CN54ENV; Biological: CN54gp140; Device: Trigrid Delivery System - Intramuscular
- Group 3: ID/EP + IM/EP (Experimental): 0.6 mg DNA-C CN54ENV, intradermally with electroporation, at Weeks 0, 4 and 8. 2 mg DNA-C CN54ENV, intramuscularly with electroporation, at Weeks 0, 4 and 8. 50 µg CN54gp140, intradermally without electroporation, at Week 20.
  Interventions: Biological: DNA-C CN54ENV; Biological: CN54gp140; Device: Trigrid Delivery System - Intramuscular; Device: Trigrid Delivery System - Intradermal

INTERVENTIONS:
Biological: DNA-C CN54ENV — DNA plasmid containing the Clade C gp140 envelope gene from HIV-1 isolate CN54
Biological: CN54gp140 — Recombinant protein expressed from the Clade C gp140 envelope gene from HIV-1 isolate CN54
Device: Trigrid Delivery System - Intramuscular — Electroporation
  Other Names: TDS-IM
  Arms: Group 2: ID + IM/EP; Group 3: ID/EP + IM/EP
Device: Trigrid Delivery System - Intradermal — Electroporation
  Other Names: TDS-ID
  Arms: Group 1: ID/EP + IM; Group 3: ID/EP + IM/EP

SUMMARY:
CUTHIVAC002 is a randomised Phase I study aimed at exploring the safety and immunogenicity of two different modes of delivery of a deoxyribonucleic acid (DNA) vaccine (DNA-C CN54ENV) via combined intramuscular and intradermal methods with and without electroporation, and boosted with recombinant HIV CN54gp140 administered by intradermal injection in healthy volunteers.

The aim of this study is to identify optimal DNA delivery conditions for promoting enhanced antibody responses to boosting with recombinant protein by the intradermal method.

DETAILED DESCRIPTION:
CUTHIVAC002 is a randomised Phase I study in healthy volunteers, aimed at exploring the safety and immunogenicity of two different modes of delivery of a deoxyribonucleic acid (DNA) HIV vaccine via combined intramuscular and intradermal methods with and without electroporation (EP), and boosted with recombinant HIV protein vaccine administered by intradermal injection without EP.

The aim of this study is to identify optimal DNA delivery conditions for promoting enhanced antibody responses to boosting with recombinant protein by the intradermal route. Healthy male and female volunteers aged 18 to 50 years old, who are at low risk of HIV infection, are to be recruited. The participants will be divided into 3 groups:

Group 1:

Participants will receive 1 x 0.15 ml (0.6 mg) DNA intradermal injections into the upper arm with EP and 1 x 0.5 ml (2 mg) intramuscular injection into the upper thigh without EP at Weeks 0, 4 & 8. And also 1 x 0.1 ml (50 μg) HIV recombinant protein by intradermal injection into the upper arm at Week 20 (final vaccination).

Group 2:

Participants will receive 1 x 0.15 ml (0.6 mg) DNA intradermal injections into the upper arm without EP and 1 x 0.5 ml (2 mg) intramuscular injection into the upper thigh with EP at weeks 0, 4 & 8. And also 1 x 0.1 ml (50 μg) HIV recombinant protein by intradermal injection into the upper arm at Week 20 (final vaccination).

Group 3:

Participants will receive 1 x 0.15 ml (0.6 mg) of DNA of intradermal injections into the upper arm with EP and 1 x 0.5 ml (2 mg) intramuscular injection into the upper thigh with EP at weeks 0, 4 & 8. And also 1 x 0.1 ml (50 μg) HIV recombinant protein by intradermal injection into the upper arm at Week 20 (final vaccination).

The investigators aim to have 8 participants complete the study in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 18 and 50 years on the day of screening
2. BMI between 18-30
3. Available for follow-up for the duration of the study (~5 months from screening)
4. Willing and able to give written informed consent
5. At low risk of HIV and willing to remain so for the duration of the study defined as:

   * no history of injecting drug use in the previous ten years
   * no gonorrhoea or syphilis in the last six months
   * no high risk partner (e.g. injecting drug use, HIV positive partner) either currently or within the past six months
   * no unprotected anal intercourse in the last six months, outside a relationship with a regular partner known to be HIV negative
   * no unprotected vaginal intercourse in the last six months outside a relationship with a regular known/presumed HIV negative partner
6. Willing to undergo a HIV test
7. Willing to undergo a genital infection screen
8. Must agree to require male sexual partner to use condoms, from at least 14 days before the first vaccination until at least 14 days after the last
9. If heterosexually active female capable of becoming pregnant, must (in addition to requiring male partner to use condoms) agree to use hormonal contraception, or to complete abstinence, from at least 14 days before the first vaccination until at least 14 days after the last. [Note: Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal, and IUD/IUS, are not acceptable methods of contraception.] If sexually active male, must agree to use condoms from the day of first vaccination until at least 14 days after the last. [Note: Additional use of an effective method of contraception is recommended for any non-pregnant female partner over the same period.]
10. Agree to abstain from donating blood for three months after the end of their participation in the trial, or longer if necessary
11. Registered with a GP for at least the past three months
12. Entered and clearance obtained from The Over-volunteering Prevention System (TOPS) database.

Exclusion Criteria:

1. Pregnant or lactating
2. History of cardiac arrhythmia or palpitations [e.g., supraventricular tachycardia, atrial fibrillation, frequent ectopy, or sinus bradycardia prior to study entry (sinus arrhythmia is not excluded)
3. History of syncope or fainting episodes within 1 year of study entry
4. History of grand-mal epilepsy, seizure disorder or any history of prior seizure
5. Individuals in which a skin-fold measurement (cutaneous and subcutaneous tissue) of the upper right or left thigh exceeds 40 mm
6. Clinically relevant abnormality on history or examination
7. Known hypersensitivity to any component of the vaccine formulations used in this trial, or have severe or multiple allergies to drugs or pharmaceutical agents
8. History of severe local or general reaction to vaccination defined as

   * local: extensive, indurated redness and swelling involving most of the antero-lateral thigh or the major circumference of the arm, not resolving within 72 hours
   * general: fever ≥39.5 °C within 48 hours; anaphylaxis; bronchospasm; laryngeal oedema; collapse; convulsions or encephalopathy within 72 hours
9. Receipt of live attenuated vaccine or HIV envelope components within 60 days or other vaccines within 14 days of enrolment
10. Receipt of an experimental vaccine containing HIV envelope components at any time in the past
11. Receipt of blood products or immunoglobulin within 4 months of screening
12. Participation in another trial of a medicinal product, completed less than 30 days prior to enrolment.
13. HIV 1 or 2 positive or indeterminate on screening.
14. Positive for hepatitis B surface antigen, hepatitis C antibody or serology indicating active syphilis requiring treatment
15. Grade 1 or above routine laboratory parameters. Hyperbilirubinaemia to be considered an exclusion criterion only when confirmed to be conjugated bilirubinaemia
16. Current use of any electronic stimulation device, such as cardiac demand pacemakers, automatic implantable cardiac defibrillator, nerve stimulators, or deep brain stimulators.
17. Presence of any surgical or traumatic metal implants at the sites of administration
18. Unable to read and speak English to a fluency level adequate for the full comprehension of procedures required in participation and consent.
19. Women with a history of toxic shock syndrome.
20. Women using an intrauterine device for contraception (as incompatible with softcup sampling)
21. Unlikely to comply with protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Lewis, MD, Principal Investigator — Imperial College London
Locations (1):
- NIHR/Wellcome Trust Imperial Clinical Research Facility, Hammersmith Hospital, Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers were recruited
Pre-assignment Details: All enrolled participants received at least one vaccination.
Period: Overall Study
Arm/Group | Group 1: ID/EP + IM | Group 2: ID + IM/EP | Group 3: ID/EP + IM/EP
Started | 9 | 8 | 11
Completed | 8 | 8 | 8
Not Completed | 1 | 0 | 3
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Population does not include replacement subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: ID/EP + IM | Group 2: ID + IM/EP | Group 3: ID/EP + IM/EP | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Median (Inter-Quartile Range); unit: years] — No age was recorded for the 4 replacement patients
  years | 31 [25 to 34] | 27 [23 to 43] | 22 [21 to 47] | 27 [22 to 43]
Sex: Female, Male [Count of Participants; unit: Participants] — No gender data were recorded for the 4 replacement patients
  Participants
    Female | 2 | 2 | 2 | 6
    Male | 6 | 6 | 6 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White British | 6 | 5 | 6 | 17
  Other White | 1 | 0 | 2 | 3
  Other | 1 | 3 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8 | 8 | 8 | 24
Body weight [Median (Inter-Quartile Range); unit: kilograms] | 82 [76 to 85] | 62 [57 to 75] | 73 [67 to 83] | 75 [66 to 83]
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kilograms per square metre] | 24 [23 to 26] | 21 [20 to 24] | 25 [23 to 27] | 24 [21 to 25]

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint
Description: Number of participants experiencing a Grade 3 or above solicited local, systemic or laboratory adverse event, or any grade of adverse event leading to a clinical decision to discontinue immunizations, or any grade of unsolicited adverse event with onset within 7 days of immunization
Time Frame: From first dose until up to Week 22
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ID/EP + IM | Group 2: ID + IM/EP | Group 3: ID/EP + IM/EP
Number analyzed (Participants) | 9 | 8 | 11
Participants | 7 | 8 | 10
Statistical Analysis 1: Comparison: Group 1: ID/EP + IM vs Group 2: ID + IM/EP vs Group 3: ID/EP + IM/EP; The proportions of subjects with primary safety outcomes were compared in a pairwise manner between the three randomised groups, using Fisher's exact tests; Test type: Other — Inequality test; p > 0.05, Fisher Exact

2. Primary Outcome: Primary Immunogenicity
Description: Magnitude of antigen-specific systemic IgG antibody binding responses (ng/mL) to CN54gp140
Time Frame: Week 22
Population: All enrolled participants
Measure: Median (Inter-Quartile Range); unit: nanograms per millilitre
Groups:
- Group 1: ID/EP + IM: 0.6 mg DNA-C CN54ENV, intradermally with electroporation, at Weeks 0, 4 and 8. 2 mg DNA-C CN54ENV, intramuscularly without electroporation, at Weeks 0, 4 and 8.
  50 µg CN54gp140, intradermally without electroporation, at Week 20.
  DNA-C CN54ENV: DNA plasmid containing the Clade C gp140 envelope gene from HIV-1 isolate CN54
  CN54gp140: Recombinant protein expressed from the Clade C gp140 envelope gene from HIV-1 isolate CN54
  Trigrid Delivery System - Intradermal: Electroporation
- Group 2: ID + IM/EP: 0.6 mg DNA-C CN54ENV, intradermally without electroporation, at Weeks 0, 4 and 8.
  2 mg DNA-C CN54ENV, intramuscularly with electroporation, at Weeks 0, 4 and 8. 50 µg CN54gp140, intradermally without electroporation, at Week 20.
  DNA-C CN54ENV: DNA plasmid containing the Clade C gp140 envelope gene from HIV-1 isolate CN54
  CN54gp140: Recombinant protein expressed from the Clade C gp140 envelope gene from HIV-1 isolate CN54
  Trigrid Delivery System - Intramuscular: Electroporation
Arm/Group | Group 1: ID/EP + IM | Group 2: ID + IM/EP | Group 3: ID/EP + IM/EP
Number analyzed (Participants) | 9 | 8 | 11
nanograms per millilitre | 13934 [9884 to 38050] | 11292 [9608 to 15568] | 31418 [6304 to 128259]
Statistical Analysis 1: Comparison: Group 1: ID/EP + IM vs Group 2: ID + IM/EP vs Group 3: ID/EP + IM/EP; Kruskal-Wallis test with Dunn's correction for multiple comparisons to compare the levels of antigen-specific serum IgG in the three groups at Week 22; Test type: Other — Inequality test; p > 0.05, Kruskal-Wallis; Kruskal-Wallis test with Dunn's correction for multiple comparisons

3. Secondary Outcome: Adverse Event Local to the Injection Sites, Starting Within 7 Days of Injection
Description: Number of participants experiencing an adverse event local to the injection sites, starting within 7 days of injection
Time Frame: 7 days after injection
Population: Population does not include replacement participants
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ID/EP + IM | Group 2: ID + IM/EP | Group 3: ID/EP + IM/EP
Number analyzed (Participants) | 8 | 8 | 8
Participants | 8 | 8 | 8

ADVERSE EVENTS:
Time Frame: Week 0 to Week 22
Arm/Group | Group 1: ID/EP + IM | Group 2: ID + IM/EP | Group 3: ID/EP + IM/EP
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 1/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: ID/EP + IM (N=9) | Group 2: ID + IM/EP (N=8) | Group 3: ID/EP + IM/EP (N=11)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Occurred 5 months after the affected subject's final vaccination
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: ID/EP + IM (N=9) | Group 2: ID + IM/EP (N=8) | Group 3: ID/EP + IM/EP (N=11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | NA | NA | 1 (1)
Fatigue (General disorders) | NA | NA | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT02589795/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT02589795/SAP_001.pdf